CLINICAL TRIAL: NCT01912339
Title: Minimally Invasive Prostatic Vapor Ablation - Multicenter, Controlled Study for the Treatment of BPH (Rezūm II)
Brief Title: Safety and Efficacy Study for the Treatment of BPH (Enlarged Prostate)
Acronym: REZUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2105-001
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptom
Keywords: Hyperplasia; Retention; Prostate
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Hyperplasia | interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Treatment: Rezūm System
  Interventions: Device: Rezum System
- Control (Other): Control: Rigid Cystoscopy
  Interventions: Procedure: Rigid Cystoscopy

INTERVENTIONS:
Device: Rezum System — The Rezūm System uses sterile water vapor (steam) to treat BPH by delivering targeted, controlled doses of stored thermal energy directly to the transition zone of the prostate gland.
  A narrow sheath, similar in shape and size to a cystoscope, is inserted transurethrally and positioned within the prostatic urethra between the bladder neck and the verumontanum.
  A thin needle is deployed through the urethra into the transition zone, and a very short (8-10 second) treatment of water vapor is delivered directly into the hyperplastic tissue and immediately disperses through the tissue interstices.
  Upon contact with the tissue, the vapor condenses, or phase shifts, into its liquid state, releasing the stored thermal energy contained within the vapor. This thermal energy is released directly against the walls of the tissue cells within the treatment zone, gently and immediately denaturing the cell membranes, thereby causing instantaneous cell death.
  Arms: Treatment
Procedure: Rigid Cystoscopy — Endoscopy of the urinary bladder via the urethra.
  Other Names: Cystoscopy
  Arms: Control

SUMMARY:
To evaluate the safety and efficacy of the Rezūm System and assess its effect on urinary symptoms secondary to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This study is a prospective, controlled, randomized single blind clinical trial of subjects with benign prostatic hyperplasia, which will allow for an interim analysis for sample size adjustment. Subjects first will be randomized in a 2:1 proportion in favor of the Treatment arm. Subjects in the Control arm will be allowed to crossover to have the Rezūm treatment after the 3-month follow-up examination.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects > 50 years of age who have symptomatic BPH.
2. International Prostate Symptom Score (IPSS) score ≥ 13.
3. Peak urinary flow rate (Qmax): ≥ 5ml/sec to ≤ 15 ml/sec with minimum voided volume of ≥ 125 ml.
4. Post-void residual (PVR) ≤250 ml.
5. Prostate volume > 30 and ≤ 80 gm.

Exclusion Criteria:

1. History of clinically significant congestive heart failure (i.e. NYHA Class III and IV).
2. History of diabetes not controlled by a stable dose of medication over the past three months. Patients with a Hemoglobin A1c that is <8.0% are allowed.
3. History of significant respiratory disease where hospitalization for the disease is required.
4. History of immunosuppressive conditions (e.g., AIDS, post-transplant).
5. Cardiac arrhythmias that are not controlled by medication or medical device.
6. An episode of unstable angina pectoris, a myocardial infarction, transient ischemic attack, or a cerebrovascular accident within the past six months.
7. Any significant medical history that would pose an unreasonable risk or make the subject unsuitable for the study.
8. Presence of a penile implant or stent(s) in the urethra or prostate.
9. Any prior invasive prostate intervention (e.g., radio frequency (RF) ablation, balloon, microwave, or laser) or other surgical interventions of the prostate.
10. Currently enrolled in any other pre-approval investigational study in the USA (does not apply to long-term post-market studies unless these studies might clinically interfere with the current study endpoints (e.g., limit use of study-required medication, etc.)).
11. History of confirmed malignancy or cancer of prostate or bladder, however, high grade PIN is acceptable.
12. History of cancer in non-genitourinary system that is not considered cured (except basal cell or squamous cell carcinoma of the skin). A potential participant is considered cured if there has been no evidence of cancer within five years of randomization.
13. Previous pelvic irradiation or radical pelvic surgery.
14. Diagnosed with active Lyme Disease (borreliosis).
15. PSA > 10 ng/ml unless prostate cancer is ruled out by biopsy. If PSA is > 2.5 ng/ml and ≤ 10 ng/ml with free PSA <25%, prostate cancer for the subject must be/had been ruled out through a negative biopsy prior to enrollment.
16. Has undergone prostate biopsy within 60 days prior to treatment date or has an imminent need for surgery.
17. Previous rectal surgery (other than hemorrhoidectomy) or known history of rectal disease.
18. Active urinary tract infection by culture within 7 days of treatment or two documented independent urinary tract infections of any type in the past 6 months.
19. Verified bacterial prostatitis within last 12 months documented by culture or non-bacterial prostatitis within the last 5 years.
20. Active or history of epididymitis within the past 3 months.
21. Neurogenic bladder, sphincter abnormalities, or poor detrusor muscle function.
22. Diagnosed or suspected primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function, sphincter function or poor detrusor muscle function.
23. Urethral strictures, bladder neck contracture, unusual anatomy or muscle spasms that would prevent the introduction and use of the device.
24. Diagnosed bladder, urethral or ureteral stones or active stone passage in the past 6 months. Stones that are known to be in the kidney and have been stable for a period exceeding 3 months are permissible.
25. Post-void residual (PVR) > 250 ml.
26. Diagnosed or suspected bleeding disorder, or coagulopathies.
27. Use of antiplatelet or anticoagulant medication except low dose aspirin (≤81 mg/day) within 10 days prior to treatment.
28. Visible hematuria with subject urine sample without a known contributing factor.
29. Subject interested in maintaining fertility.
30. Use of beta-blockers, anticonvulsants, and antispasmodics where the dose is not stable. (Stable dose is defined as having the same medication and dose in the last six months).
31. At the time of baseline assessment, in the absence of a qualifying exception, subjects who are using or have used the following medications, and are unable or unwilling to discontinue using these medications for the prescribed washout period:

    1. Use of antihistamines within 1 week of treatment unless there is documented evidence of stable dosing for last 6 months (no dose changes).
    2. Use of the alpha blockers for BPH and anticholinergics or cholinergics (except for topical anti cholinergic eye drops), or within 4 weeks of baseline assessment.
    3. Use of Type II, 5-alpha reductase inhibitor (e.g., finasteride (Proscar, Propecia) within 3 months of baseline assessment.
    4. Use of a dual 5-alpha reductase inhibitor (e.g., dutasteride (Avodart)) within 6 months of baseline assessment.
    5. Use of estrogen, drug-producing androgen suppression, or anabolic steroids within 3 months of baseline assessment.
    6. Use of daily dose PD5 Inhibitors (e.g.Viagra, Levitra or Cialis) within 4 weeks of baseline assessment.
32. Subjects who have had an incidence of spontaneous urinary retention either treated with indwelling transurethral catheter or suprapubic catheter six months prior to baseline. A provoked episode now resolved is still admissible.
33. Compromised renal function defined as serum creatinine > 2.0 mg/dl.
34. Inability to provide a legally effective Informed Consent Form (ICF) and/or comply with all the required follow-up requirements.
35. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affect the ability to complete the study quality of life questionnaires.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roehrborn, MD, Principal Investigator — UT Southwestern; Kevin McVary, MD, Principal Investigator — Southern Illinois University
Locations (15):
- United States (15):
  - Arizona Institute of Urology, Tucson, Arizona
  - Urology Associates of Denver, Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Southern Illinois University, Springfield, Illinois
  - Chesapeake Urology, Towson, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Metro Urology, Woodbury, Minnesota
  - Manhattan Medical Research, New York, New York
  - The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Texas Urology, Carrollton, Texas
  - UT Southwestern, Dallas, Texas
  - Urology of San Antonio, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Rezum is a transurethral needle ablation procedure to treat BPH that can be performed in a clinic or out-patient setting. Rezum uses the stored thermal energy in water vapor (steam) to treat the extra prostate tissue that is causing symptoms such as frequency, urgency, irregular flow, weak stream, straining and getting up at night to urinate.
  Inside a hand-held device, radiofrequency energy is applied to a few drops of water to create vapor (steam). The water vapor is injected into the prostate tissue that is blocking the flow of urine from the bladder, where it immediately turns back to water, releasing the energy stored in the vapor into the cell membranes. At this point, the cells are gently and immediately damaged, causing cell death. Over time, your body will absorb the treated tissue through its natural healing response.
- Crossover of Control Subjects: Subjects randomized to the control group will be offered the option to receive the Rezum treatment after the 3 month follow-up visit evaluations are completed. Subjects must decide to cross over by the end of the 6 month follow-up visit.
Period: Blinded (0 to 3 Months)
Arm/Group | Treatment | Control | Crossover of Control Subjects
Started | 136 | 61 | 0
Completed | 134 | 61 | 0
Not Completed | 2 | 0 | 0
Not completed — Declined to participate | 1 | 0 | 0
Not completed — Open Prostatectomy | 1 | 0 | 0
Period: Unblinded (3 to 6 Months/Crossover)
Arm/Group | Treatment | Control | Crossover of Control Subjects
Started | 134 | 61 | 0
Completed | 133 (Still in study) | 61 (Of the 61 subjects, there were 53 crossover subjects and 8 that completed their study participation.) | 0 (Still in study)
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Unblinded (6 Months/Crossover to 5 Yrs)
Arm/Group | Treatment | Control | Crossover of Control Subjects
Started | 133 | 0 (All subjects for the control group either completed study or crossed over.) | 53 (Control subjects that have crossed over.)
Completed | 0 | 0 | 0
Not Completed | 133 | 0 | 53
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Missed Visit | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — BPH Medication | 1 | 0 | 0
Not completed — TURP/Laser | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Subject started on Cialis | 0 | 0 | 1
Not completed — Had PVP - Prostate laser surgery | 0 | 0 | 1
Not completed — Still in Study | 120 | 0 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 136 | 61 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 36 | 120
  >=65 years | 52 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.1) | 62.9 (7.0) | 62.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 136 | 61 | 197
Region of Enrollment [Number; unit: participants]
  United States | 136 | 61 | 197

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Change From Baseline in the International Prostate Symptom Score (IPSS) at 3 Month Follow-Up
Description: Comparison of the change in BPH symptoms as measured by IPSS change between the Treatment and Control arm at 3 months post-treatment. The IPSS is a well-validated, highly reliable and responsive American Urological Association symptom score (AUASS) assessment to identify the severity of BPH Symptoms. The first seven questions of the IPSS Questionnaire address frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying and urgency each on a scale of 0 to 5. The total score, summed across the seven items measured, ranges from 0 (no symptoms) to 35 (most severe symptoms).
Time Frame: 3 Month Follow-up Visit
Population: Intention to Treat population (ITT)
Measure: Mean (95% Confidence Interval); unit: Cange in IPSS score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 136 | 61
Cange in IPSS score | -11.2 [-12.5 to -9.9] | -4.3 [-6.1 to -2.5]

2. Primary Outcome: Safety: Device Related Serious Complications
Description: This safety endpoint will be to demonstrate that the composite observed rate of post-procedure device related serious complications in the Treatment Arm are is less than or equal to 12% at 3 months.
  Composite device related serious complications for this endpoint are 1) De Novo (new) severe urinary retention lasting more than 21 consecutive days post treatment, 2) Device related formation of fistula between the rectum and urethra, and 3) device perforation of the rectum or GI tract. Twelve percent was a pre-specified performance goal for the safety endpoint.
Time Frame: 3 Months
Population: Intention to Treat population (ITT) for treatment arm subjects only. Control subjects did not undergo a treatment procedure so they were not assessed for this endpoint.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 136 | 0
Participants | 1 [0 to 4.6] |

3. Secondary Outcome: Responders at 3 Months
Description: Number of subjects with a greater than or equal to 30% improvement (reduction) in the International Prostate Symptom score (IPSS) at 3 months compared to baseline.
Time Frame: 3 Months
Population: Intention to Treat population (ITT)
Measure: Number; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 136 | 61
Participants | 106 | 21

4. Secondary Outcome: Responders at 6 Months
Description: Number of subjects with a greater than or equal to 30% improvement (reduction) in the International Prostate Symptom score (IPSS) at 6 months compared to baseline.
Time Frame: 6 Months
Population: Intention to Treat population (ITT) for treatment subjects only. Control subjects randomized follow-up concluded at 3 months.
Measure: Number; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 136 | 0
Participants | 102 |

5. Secondary Outcome: Responders at 12 Months
Description: Number of subjects with a greater than or equal to 30% improvement (reduction) in the International Prostate Symptom score (IPSS) at 12 months compared to baseline.
Time Frame: 12 Months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 136 | 0
Participants | 104 |

ADVERSE EVENTS:
Time Frame: 1 year,10 months
Description: Within 1 year and 10 months of first enrollment (average Treatment group follow-up of 16.4 months, average Control group follow-up of 4.7 months). Procedure relatedness was adjudicated by an independent Clinical Events Committee (CEC).
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 18/136 | 4/61
Other Adverse Events (participants affected / at risk) | 66/136 | 4/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=136) | Control (N=61)
Nausea (General disorders) | 1 (1) | 0 (0) — Related to procedure
Vomiting (General disorders) | 1 (1) | 0 (0) — Related to procedure
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) — Related to procedure
UTI, Culture Proven (Renal and urinary disorders) | 1 (1) | 0 (0) — Not related to procedure
Bowel Obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0) — Not related to procedure
Injury, other (fractured ribs) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to procedure
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — Not related to procedure
Cancer, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Not related to procedure
Hemorrhoids (Vascular disorders) | 1 (1) | 0 (0) — Not related to procedure
Infection (other than UTI) (Infections and infestations) | 1 (1) | 1 (1) — Not related to procedure
Other - Atherosclerotic Artery Disease (Vascular disorders) | 1 (1) | 0 (0) — Not related to procedure
Other, Broken Right Thumb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to procedure
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Not related to procedure
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) — Not related to procedure
Spinal Stenosis (Nervous system disorders) | 1 (1) | 0 (0) — Not related to procedure
Syncope (General disorders) | 1 (1) | 1 (1) — Not related to procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=136) | Control (N=61)
Dysuria (Renal and urinary disorders) | 23 (24) | 1 (1)
Hematuria, Gross (Renal and urinary disorders) | 17 (17) | 0 (0)
Hematospermia (Reproductive system and breast disorders) | 10 (10) | 0 (0)
Urinary, Frequency (Renal and urinary disorders) | 9 (9) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 8 (8) | 1 (1)

LIMITATIONS AND CAVEATS:
All adverse events reported, including those not related to the Rezum procedure. Events related to the procedure are summarized in McVary 2016 (see "Publications automatically indexed to this study").

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less